CLINICAL TRIAL: NCT03005405
Title: Cost-efficacy and Applicability of the Treatment of Moderate Caries Using Sealants as an Alternative to the Restorations on Occlusal Surfaces of Deciduous Teeth: a Randomized Controlled Trial
Brief Title: Cost-efficacy of Sealing Moderate Caries Lesions in Occlusal Surfaces of Primary Molars
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Mariana Minatel Braga, PhD, Associate Professor, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SEALANT-CARDEC02
Record Dates: First submitted 2016-08-17; First posted 2016-12-29 (Estimated); Last update posted 2018-03-22 (Actual); Status verified 2018-03

CONDITIONS: Dental Caries
Keywords: Dental Caries; Primary tooth; Ionomer Sealants; Glass Ionomer Restoration
MeSH Terms: conditions — Dental Caries | interventions — Glass Ionomer Cements

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- restoration - control (Active Comparator): Restoration
  Interventions: Procedure: Ionomer Restoration (control); Procedure: Oral hygiene orientation and professional fluoride application
- sealant - test (Experimental): Sealant
  Interventions: Procedure: Ionomer Sealant (test); Procedure: Oral hygiene orientation and professional fluoride application

INTERVENTIONS:
Procedure: Ionomer Restoration (control) — Restoration of moderate caries lesions after partial caries removal using high viscosity glass ionomer cements
  Other Names: glass ionomer cement, restoration
  Arms: restoration - control
Procedure: Ionomer Sealant (test) — Sealing of moderate caries lesions without any caries removal or cavity opening.
  Other Names: glass ionomer cement, sealant
  Arms: sealant - test
Procedure: Oral hygiene orientation and professional fluoride application — Oral hygiene orientation and professional fluoride application

SUMMARY:
This protocol aims to assess the cost-efficacy and applicability of the treatment of lesions moderate caries using sealants as an alternative to the restorations on occlusal surfaces of deciduous teeth. Initially, a non-inferiority study was designed in order to verify if sealing could be non-inferior than restoration. In this case, it could be preferable since it is less invasive. Therefore, cost will be put forward into the analysis considering even reintervention during the follow-ups (cost-efficacy analyses). Finally, the acceptability could be another differential point between treatments.

DETAILED DESCRIPTION:
This study aims to evaluate the cost-efficacy and applicability of the treatment of lesions moderate caries using sealants as an alternative to the restorations on occlusal surfaces of deciduous teeth. 96 children aged 3-6 years will be selected. Children must have at least one occlusal surface classified as scores 3 or 4 of International Caries Detection and Assessment System (ICDAS). Children will be randomly allocated according to the treatment: glass ionomer sealant and restoration with glass ionomer. After treatment, teeth will be assessed clinically after 6, 12, 18 and 24 months by trained and blinded examiners regarding the treatment received. The need of reintervention initially treated, either by failures that require repeating of the same procedure or for progression of caries lesions will be considered as primary outcomes. The secondary outcomes will be the chil's acceptability to the treatment.

ELIGIBILITY:
Inclusion Criteria:

They will be included in this study children:

* aged 3 years and 6 years and 11 months;
* With complete primary dentition;
* Who have at least one active caries lesion score 3 or 4 ICDAS, in the occlusal molars surfaces.
* Who have assented to participate and whose parents have consented to their participation by signing the Instrument of Consent.

Exclusion Criteria:

* who have medical and / or behavioral conditions that require special considerations regarding handling / treatment;
* who are involved in other research that may impact on this study;
* whose parents that not agree in participate.

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 96 (Estimated)
Dates: Start 2015-02; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Need of reintervention | 24 months
  Need of reintervention will be considered as all failures after initial treatment that demand repair and/or caries progression associated to the treated lesion at baseline.
  After cleaning, It will be analyzed the clinical evaluation of restorations and sealants, will be assessed the presence of caries lesions in dentin and / or evolution of ICDAS scores and if will be necessary other types of treatment, such as endodontics and extraction of teeth included.

SECONDARY OUTCOMES:
Child's reported discomfort | 1st day
  The discomfort will be an outcome collected right after the end of treatment, using Wong baker scale
Duration of treatments | 1st day
  Time spent in interventions will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Mariana M Braga, PhD, Principal Investigator — University of Sao Paulo
Locations (1):
- University of São Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Publication of all results, accessibility to data if necessary